CLINICAL TRIAL: NCT03006536
Title: Low-Intensity Extracorporeal Shock Wave Treatment for Erectile Dysfunction: A Randomized, Controlled, Double Blind Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Nessn Azawi, Chief Urologist, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJ-590
Record Dates: First submitted 2016-12-26; First posted 2016-12-30 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Li-ESWT (Experimental): Participants will undergo 6 treatment sessions 2/week with 1 week pause with the Duolith® SD1 machine (Storz, Tägerwilen, Switzerland) according to the company's instructions
  Interventions: Device: Li-ESWT
- Sham (Sham Comparator): Participants will undergo 6 treatment sessions 2/week with 1 week pause with the Duolith® SD1 machine (Storz, Tägerwilen, Switzerland) according to the company's instructions
  Interventions: Device: Li-ESWT

INTERVENTIONS:
Device: Li-ESWT — Participants will undergo 6 treatment sessions 2/week with 1 week pause with the Duolith® SD1 machine (Storz, Tägerwilen, Switzerland) according to the company's instructions

SUMMARY:
The proposed mechanism of action for LI-ESWT in ED is that it improves endothelial function and triggers angiogenesis through induction of local growth factors and endothelial nitric oxide synthase. The literature generally confirms that LI-ESWT is safe and cohort studies investigating the clinical effects have been encouraging. Meanwhile, randomized trials have shown contradictory results. Thus, a randomized trial in 67 PDE5-I responders showed statistically greater improvements in the Erectile Function Domain of the International Index of Erectile Function (IIEF) with active LI-ESWT treatment compared to a sham treatment (p=0.032).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* A history of erectile dysfunction for >6 months
* IIEF-ED score < 25
* In a stable heterosexual relationship for at least 6 months
* Willingness to attempt sexual intercourse at least twice per week during the study and follow-up

Exclusion Criteria:

* Psychogenic ED as assessed by a standardized interview (attachment 2)
* Known psychiatric illness
* Neurological disease (including Parkinson's disease, Multiple sclerosis, spinal cord injury, and a history of stroke)
* Traumatic nerve injury
* Previous pelvic surgery or radiation
* Heart disease in the form of unstable angina, NYHA class >II heart failure, uncontrolled arrhythmia, or significantly symptomatic and/or severe valvular disease
* Endocrine disease including hypogonadism (total testosterone <12 nmol/l)
* Insulin dependent or uncontrolled diabetes mellitus
* Dependence on erectogenic aids other than PDE5-Inhibitors
* Use of medications which have been shown to interfere with erections
* Use of anticoagulant medications other than low dose aspirin
* Active cancer
* A diagnoses of Peyronie's disease and/or prior occurrence of priapism
* Alcohol abuse (more than 21 containers of alcohol per week)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF) | 1 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Roskilde, Denmark